CLINICAL TRIAL: NCT06331377
Title: Clinical and Molecular Characteristics of Histiocytic Disorders
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 17-004541; NCI-2024-01765 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 17-004541 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2024-03-18; First posted 2024-03-26 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Histiocytic Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (1):
- Observational: Patients complete questionnaires and undergo blood and tissue sample collection. Patients' medical records are also reviewed.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study

SUMMARY:
This study is being done to collect medical and personal histories as well as a samples of blood, other body fluid and/or tumor/disease tissue for current and future research studies on histiocytic disorders.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Define molecular signature and genomic landscape of histiocytic disorders. II. Correlate genomic findings with transcriptional abnormalities. III. Identify promising prognostic alterations and potential therapeutic targets.

OUTLINE: This is an observational study.

Patients complete questionnaires and undergo blood and tissue sample collection. Patients' medical records are also reviewed.

ELIGIBILITY:
Inclusion Criteria:

* * All patients diagnosed with histiocytic disorders and age ≥1 year

Exclusion Criteria:

* * < 1 years age

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients diagnosed with histiocytic disorders
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-07-27 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Identify molecular markers | Baseline
  Biopsy samples will be analyzed for the presence of molecular markers associated with histiocytic disorders. Potential markers include BRAF V600E, cyclinD1, PD-L1, p16, and p53.6. For any test results that are actionable, patients will be notified and the results will be available in the electronic medical record.
Change in PD-L1 and T-cell Bim expression | Baseline; post-treatment (estimated up to 2 years, potentially 4 times per year)
  Blood testing will be performed for soluble PD-L1 and T-cell Bim expressions before and after radiation therapy for histiocytic disease to assess change in levels and role of immunotherapy. For any test results that are actionable, patients will be notified and the results will be available in the electronic medical record.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald S. Go, M.D., Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials